CLINICAL TRIAL: NCT03548077
Title: Harmonization Project: Men's Healthy Eating Active Living (MHEAL)
Brief Title: POWERPLAY: Promoting Men's Health at Work
Acronym: POWERPLAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Athabasca University (Other); Northern Health, British Columbia, Canada (Unknown); British Columbia Cancer Agency (Other); Canadian Cancer Society (CCS) (Other)
Responsible Party: Principal Investigator, Joan Bottorff, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 702831
Record Dates: First submitted 2018-05-24; First posted 2018-06-06 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-10

CONDITIONS: Men; Health Behavior; Health Knowledge, Attitudes, Practice; Cancer
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1; Health Behavior; Behavior; Neoplasms

STUDY DESIGN:
Intervention Model Description: Quasi-experimental, pre-post study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention group (Experimental): Powerplay, a workplace wellness program designed for male-dominated work sites, is the intervention. The program focuses on physical activity, healthy eating, mental wellness, and smoking cessation as well as promoting changes in workplace environments to support employee health and wellness. Program delivery is supported with a detailed program manual and web-based resources. More information about the intervention is available here: http://www.powerplayatwork.com/
  Interventions: Behavioral: POWERPLAY

INTERVENTIONS:
Behavioral: POWERPLAY — All men from participating worksites are invited to completed surveys prior to and following implementation of a workplace wellness program (called "POWERPLAY")

SUMMARY:
With funding from the Candian Cancer Society, the Men's Healthy Eating Active Living (MHEAL) project began the development, evaluation, and optimization of a program called POWERPLAY to promote men's health at work.

DETAILED DESCRIPTION:
The MHEAL project began November 2013 and a program (called "POWERPLAY") was developed to support men's active living and healthy eating based on a systematic review of the literature and consultations with groups of men. From 2014-2017 six male-dominated worksites in northern BC offered POWERPLAY and participated in this study. Using a quasi-experimental pre-post design as well as interviews with worksite leads, the program was demonstrated to be an effective, feasible, and acceptable approach to the promotion of modifiable behaviours known to reduce the risk of cancer among working men in northern settings, and several manuscripts were published. Furthermore, the POWERPLAY program was optimized based on feedback received to include friendly competitions, weekly motivational messages, men-friendly language/images, and pedometers, and a manual for employers and website were developed (http://www.powerplayatwork.com/). A new module to support mental well-being was created in 2017 based on a systematic review of the literature for men's mental wellness programs, consultations with men working in northern workplaces, and interviews with workplace representatives. A module to support smoking cessation module was created in 2018.

ELIGIBILITY:
Inclusion Criteria:

Men employed in participating workplaces, full-time or part-time, in any position within the organization

Exclusion Criteria:

Although females were not discouraged from participating in the POWERPLAY program, they were not included in the evaluation.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility based on self-representation of gender identity
Enrollment: 227 (Actual)
Dates: Start 2014-09-24 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Physical Activity | 6 months
  Weekly physical activity was assessed using the Godin Leisure-Time Exercise Questionnaire (Godin & Shephard, 1985).

SECONDARY OUTCOMES:
Healthy Eating | 6 months
  Self-reported servings of fruits and vegetables

CONTACTS AND LOCATIONS:
Overall Officials: Joan L Bottorff, PhD, RN, Principal Investigator — University of British Columbia
Locations (1):
- Faculty of Health and Social Development, Kelowna, British Columbia, Canada

REFERENCES:
- [Background] Bottorff JL, Seaton CL, Johnson ST, Caperchione CM, Oliffe JL, More K, Jaffer-Hirji H, Tillotson SM. An Updated Review of Interventions that Include Promotion of Physical Activity for Adult Men. Sports Med. 2015 Jun;45(6):775-800. doi: 10.1007/s40279-014-0286-3. PMID 25430599
- [Background] Caperchione CM, Sharp P, Bottorff JL, Stolp S, Oliffe JL, Johnson ST, Jones-Bricker M, Errey S, Christian H, Healy T, Medhurst K, Lamont S. The POWERPLAY workplace physical activity and nutrition intervention for men: Study protocol and baseline characteristics. Contemp Clin Trials. 2015 Sep;44:42-47. doi: 10.1016/j.cct.2015.07.013. Epub 2015 Jul 14. PMID 26187657
- [Background] Oliffe JL, Bottorff JL, Sharp P, Caperchione CM, Johnson ST, Healy T, Lamont S, Jones-Bricker M, Medhurst K, Errey S. Healthy Eating and Active Living: Rural-Based Working Men's Perspectives. Am J Mens Health. 2017 Nov;11(6):1664-1672. doi: 10.1177/1557988315619372. Epub 2015 Dec 14. PMID 26669775
- [Background] Seaton CL, Bottorff JL, Jones-Bricker M, Oliffe JL, DeLeenheer D, Medhurst K. Men's Mental Health Promotion Interventions: A Scoping Review. Am J Mens Health. 2017 Nov;11(6):1823-1837. doi: 10.1177/1557988317728353. Epub 2017 Sep 8. PMID 28884637
- [Result] Johnson ST, Stolp S, Seaton C, Sharp P, Caperchione CM, Bottorff JL, Oliffe JL, Jones-Bricker M, Lamont S, Medhurst K, Errey S, Healy T. A Men's Workplace Health Intervention: Results of the POWERPLAY Program Pilot Study. J Occup Environ Med. 2016 Aug;58(8):765-9. doi: 10.1097/JOM.0000000000000793. PMID 27281710
- [Result] Caperchione CM, Stolp S, Bottorff JL, Oliffe JL, Johnson ST, Seaton C, Sharp P, Jones-Bricker M, Lamont S, Errey S, Healy T, Medhurst K, Christian H, Klitch M. Changes in Men's Physical Activity and Healthy Eating Knowledge and Behavior as a Result of Program Exposure: Findings From the Workplace POWERPLAY Program. J Phys Act Health. 2016 Dec;13(12):1364-1371. doi: 10.1123/jpah.2016-0111. Epub 2016 Sep 6. PMID 27617968
- [Result] Seaton CL, Bottorff JL, Oliffe JL, Jones-Bricker M, Caperchione CM, Johnson ST, Sharp P. Acceptability of the POWERPLAY Program: A Workplace Health Promotion Intervention for Men. Am J Mens Health. 2017 Nov;11(6):1809-1822. doi: 10.1177/1557988317728354. Epub 2017 Sep 8. PMID 28884636
- See also: POWERPLAY program website — http://www.powerplayatwork.com/
- See also: Research project website for MHEAL — http://harmonization.ok.ubc.ca/mens-healthy-eating-active-living/